CLINICAL TRIAL: NCT00824798
Title: Gait Evaluation in Haemophiliac Patients
Acronym: GAIT_GENERAL
Status: Completed | Type: Observational
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Other Study IDs: READ-LOBET-02
Record Dates: First submitted 2009-01-16; First posted 2009-01-19 (Estimated); Last update posted 2019-07-11 (Actual); Status verified 2019-07

CONDITIONS: Hemophilia A; Hemophilia B
Keywords: gait; haemophilia; arthropathy
MeSH Terms: conditions — Hemophilia A; Hemophilia B; Joint Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- haemophiliacs A and B: haemophiliacs A and B mild, moderate or severe from 4 to 80 years old, with or without inhibitors.

SUMMARY:
Joint damage secondary to recurrent haemarthroses and chronic synovitis represents the commonest clinical manifestation of haemophilia. Incapacitating pain, loss of joint stability and mobility, axial deviation, deterioration and decreased function are the most frequent complains in patients with severe haemophilic arthropathy In this context, the purpose of our study is to examine and analyse specific changes in gait in patients suffering from haemophilic arthropathy and determine the impact on health-related quality of life in terms of conceptual components of pain and stiffness, psychosocial stress, disability, and activity limitations as recommended by the International Classification of Function (ICF) recently published by the World Health Organization.

ELIGIBILITY:
Inclusion Criteria:

* haemophilia A or B
* aged more than 4 years

Exclusion Criteria:

* impossibility to walk on a treadmill
* recent joint haemarthrosis or muscle haematoma

Ages: 5 Years to 80 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: haemophilia A or B, mild, moderate or severe.
Sampling Method: Non-Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2009-01; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
evaluate specific changes in gait in patients suffering from haemophilic arthropathy | from inclusion in the study until 1 year after inclusion

CONTACTS AND LOCATIONS:
Overall Officials: sebastien lobet, Principal Investigator — sebastien.lobet@uclouvain.be
Locations (1):
- Cliniques universitaires Saint-Luc, Brussels, Belgium

REFERENCES:
- [Result] Lobet S, Detrembleur C, Francq B, Hermans C. Natural progression of blood-induced joint damage in patients with haemophilia: clinical relevance and reproducibility of three-dimensional gait analysis. Haemophilia. 2010 Sep 1;16(5):813-21. doi: 10.1111/j.1365-2516.2010.02245.x. Epub 2010 Apr 7. PMID 20398067
- [Result] Lobet S, Hermans C, Pasta G, Detrembleur C. Body structure versus body function in haemophilia: the case of haemophilic ankle arthropathy. Haemophilia. 2011 May;17(3):508-15. doi: 10.1111/j.1365-2516.2010.02433.x. Epub 2011 Mar 4. PMID 21371180
- [Result] Lobet S, Hermans C, Bastien GJ, Massaad F, Detrembleur C. Impact of ankle osteoarthritis on the energetics and mechanics of gait: the case of hemophilic arthropathy. Clin Biomech (Bristol). 2012 Jul;27(6):625-31. doi: 10.1016/j.clinbiomech.2012.01.009. Epub 2012 Feb 29. PMID 22381586
- [Result] Lobet S, Detrembleur C, Hermans C. Impact of multiple joint impairments on the energetics and mechanics of walking in patients with haemophilia. Haemophilia. 2013 Mar;19(2):e66-72. doi: 10.1111/hae.12001. Epub 2012 Sep 9. PMID 22958138
- [Result] Lobet S, Detrembleur C, Massaad F, Hermans C. Three-dimensional gait analysis can shed new light on walking in patients with haemophilia. ScientificWorldJournal. 2013 May 13;2013:284358. doi: 10.1155/2013/284358. Print 2013. PMID 23766686